CLINICAL TRIAL: NCT00683852
Title: A Double-Blind, Placebo-Controlled Study of Aripiprazole Adjunctive to Antidepressant Therapy (ADT) Among Outpatients With Major Depressive Disorder Who Have Responded Inadequately to Prior ADT
Brief Title: A Double-Blind, Placebo-Controlled Study of Aripiprazole Adjunctive to Antidepressant Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Executive Vice Chair, Department of Psychiatry; Executive Director, Clinical Trials Network and Institute (CTNI); Director, Depression Clinical and Research Program (DCRP), Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BMS - 2008A053242
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Drug 2mg/Drug 5mg (Active Comparator): patients randomly assigned to the drug/drug sequence, the dose of aripiprazole will be 2 mg/day during the first phase of the study, and 5 mg/day in the second phase.
  Interventions: Drug: Aripiprazole 5mg; Drug: Aripiprazole 2mg
- Placebo/Drug 2mg (Active Comparator): For patients randomly assigned to the placebo/drug sequence, the dose of aripiprazole will be 2 mg/day during the second phase of the study.
  Interventions: Drug: Aripiprazole 2mg; Drug: Placebo
- Placebo/Placebo (Placebo Comparator): for patients randomly assigned to the placebo/placebo sequence, study medication will be placebo during both phases of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole 5mg — Tablet dose of aripiprazole will be 2 mg/day during the first phase (30 days) of the study, and 5 mg/day in the second phase (30 days)
  Other Names: Abilify
  Arms: Drug 2mg/Drug 5mg
Drug: Aripiprazole 2mg — For patients randomly assigned to the placebo/drug sequence, the dose of aripiprazole will be 2 mg/day during the second phase of the study (30 days)
  Other Names: Abilify
  Arms: Drug 2mg/Drug 5mg; Placebo/Drug 2mg
Drug: Placebo — for patients randomly assigned to the placebo/placebo sequence, study medication will be placebo during both phases of the study (60 days)
  Arms: Placebo/Drug 2mg; Placebo/Placebo

SUMMARY:
The purpose of this study is to determine whether a reduced dose of aripiprazole is effective in treating patients with major depressive disorder

DETAILED DESCRIPTION:
This is a 60-day, multi-center, double-blind, placebo-controlled study on the efficacy of aripiprazole (Abilify) augmentation of selective serotonin reuptake inhibitors (SSRIs) or selective serotonin norepinephrine uptake inhibitors (SNRIs) venlafaxine in patients with MDD who have responded inadequately to treatment with ADTs. The purpose of our study is to evaluate the efficacy and tolerability of low-dose (2 mg/day) aripiprazole (Abilify) as an augmentation strategy in MDD non-responding to ADT with SSRIs or the SNRI venlafaxine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to give informed consent, and/or consent obtained from a legally acceptable representative (as required by IRB/IEC), prior to the initiation of any protocol required procedures.
2. Patients must be able to understand the nature of the study, agree to comply with the prescribed dosage regimens, report for regularly scheduled office visits, and communicate to study personnel about adverse events and concomitant medication use.
3. Patients with a diagnosis of major depressive episode as defined by DSM-IV-TR criteria, based on the SCID-I/P; their major depressive episode must be deemed "valid" using the SAFER criteria interview administered by remote, independent raters.
4. Patients who have reported a history for the current depressive episode of an inadequate response to at least one and no more than three adequate antidepressant treatments. An inadequate response is defined as less than a 50% reduction in depressive symptom severity, as assessed by the MGH ATRQ administered by remote, independent raters. An adequate trial is defined as an antidepressant treatment for at least 6 weeks duration at least at a minimum dose as specified in the MGH ATRQ.
5. Patients must have a HAM-D17 ≥ 18 at the end of the screening phase to qualify for inclusion. The HAM-D17 will be administered by the study clinicians at the screening and baseline visits, and by remote, independent raters during the screening phase at the time of the SAFER interview.
6. Patients must be able to be reliably rated on the psychiatric scales required by the protocol.
7. Men and women, ages 18 to 65 Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized.

   WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea ³ 12 consecutive months; or women on hormone replacement therapy [HRT] with documented serum follicle stimulating hormone [FSH] level > 35 mIU/mL). Even women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential.

   WOCBP must have a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of investigational product.
8. Meet DSM-IV criteria (by Structured Clinical Interview for DSM-IV - SCID-I/P) for MDD, current;
9. Quick Inventory of Depressive Symptomatology - Self-Rated (QIDS-SR) (22) score of at least 16 at both screen and baseline visits;
10. Treated with an SSRI at adequate doses (defined as 20mg/day or more of fluoxetine, citalopram; paroxetine 30mg/day or more or 37.5 mg/day or more of paroxetine CR; 10 mg/day or more of escitalopram, 50mg/day or more of sertraline, and 150 mg/day or more of venlafaxine) during the current episode for at least 8 weeks, with the same, adequate dose over the last 4 weeks;
11. Between the screen and baseline visit, patients must be documented prospectively to have received a stable dose of their SSRI or venlafaxine for at least 2 weeks.

Additional criteria for defining response and non-response for patients in Phase 2 eligible for the pooling of the data with all the patients in Phase 1. Among patients pre-randomized to receive placebo in both phases or to receive placebo in Phase 1 and aripiprazole in phase 2, only those meeting non-response criteria will be added to the primary efficacy sample:

* Placebo non-responders are defined as those patients who failed to achieve a 50% decrease in their MADRS score at visit 3,
* Have a MADRS score of > 16 at visit 3

Exclusion Criteria:

1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period [and for up to 4 weeks after the last dose of investigational product].
2. WOCBP using a prohibited contraceptive method.
3. Women who are pregnant or breastfeeding.
4. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
5. Sexually active fertile men not using effective birth control if their partners are WOCBP.
6. Patients who report an inadequate response (less than 50% decrease in depressive symptom severity) to more than two adequate trials of antidepressant treatments during the current depressive episode (including monotherapy treatment and distinct combination regimens) at a therapeutic dose (as defined by the ATRQ) and for an adequate duration (minimum six weeks for any monotherapy).
7. Patients who report treatment with adjunctive antipsychotic medication with an antidepressant for a minimum of two weeks during the current depressive episode.
8. Patients with a current need for involuntary commitment or who have been hospitalized within four weeks of the Screening Visit for the current major depressive episode.
9. Patients who have received ECT during the current episode.
10. Patients who have a current Axis I diagnosis of:

    1. Delirium, dementia, amnestic, or other cognitive disorder;
    2. Schizophrenia or other psychotic disorder, based on the SCID-I/P;
    3. Bipolar I or II disorder, based on the SCID-I/P;
11. Patients with a clinically significant Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder.
12. Patients experiencing hallucinations, delusions, or any psychotic symptomatology in the current depressive episode.
13. Patients who have met DSM-IV-TR criteria for any significant substance use disorder within the past six months, based on the SCID-I/P.
14. Patients receiving new onset psychotherapy within 6 weeks of screening, or at any time during participation in the trial.
15. Patients who have been previously randomized in an aripiprazole clinical trial (lifetime).
16. Patients who have participated in any clinical trial with an investigational drug or device within the past month.
17. Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease;
18. Patients who, in the investigator's judgment represent a significant risk of committing suicide during the course of the trial based on history or evaluation of current mental status
19. Patients who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the course of the trial
20. Patients with thyroid pathology (unless condition has been stabilized with medications for at least the past three months)
21. Patients with a lifetime history of neuroleptic malignant syndrome or serotonin syndrome
22. Patients with a significant history of a seizure disorder
23. Patients with detectable levels of cocaine, heroin or opioids in the urine drug screen
24. Diastolic blood pressure > 105 mmHg
25. Any signs or symptoms that in the investigator's judgment are medically significant, in that it would impact the patients safety.

    1. Patients who are known to be allergic or hypersensitive to aripiprazole or other dihydrocarbostyrils (e.g. carteolol, vesnarinone, and cilostazol)
    2. Patients previously treated with and not responding to aripiprazole
    3. Monoamine oxidase inhibitors (e.g., Nardil, phenelzine, Parnate, tranylcypromine, Marplan, isocarboxazid) treatment within the two weeks prior to enrollment
    4. Patients who would likely require prohibited concomitant medication during the trial
    5. Prisoners or subjects who are involuntarily incarcerated
    6. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
    7. Patients who no longer meet DSM-IV criteria for MDD during the baseline visit;
    8. Patients who demonstrate a greater than 25% decrease in depressive symptoms as reflected by the QIDS-SR or HAM-D17 total score from screen visit to baseline visit;
    9. Patients with a history of antidepressant-induced hypomania.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Marcus RN, McQuade RD, Carson WH, Hennicken D, Fava M, Simon JS, Trivedi MH, Thase ME, Berman RM. The efficacy and safety of aripiprazole as adjunctive therapy in major depressive disorder: a second multicenter, randomized, double-blind, placebo-controlled study. J Clin Psychopharmacol. 2008 Apr;28(2):156-65. doi: 10.1097/JCP.0b013e31816774f9. PMID 18344725
- [Background] Berman RM, Marcus RN, Swanink R, McQuade RD, Carson WH, Corey-Lisle PK, Khan A. The efficacy and safety of aripiprazole as adjunctive therapy in major depressive disorder: a multicenter, randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2007 Jun;68(6):843-53. doi: 10.4088/jcp.v68n0604. PMID 17592907
- [Result] Fava M, Mischoulon D, Iosifescu D, Witte J, Pencina M, Flynn M, Harper L, Levy M, Rickels K, Pollack M. A double-blind, placebo-controlled study of aripiprazole adjunctive to antidepressant therapy among depressed outpatients with inadequate response to prior antidepressant therapy (ADAPT-A Study). Psychother Psychosom. 2012;81(2):87-97. doi: 10.1159/000332050. Epub 2012 Jan 25. PMID 22286203
- [Derived] Mischoulon D, Witte J, Levy M, Papakostas GI, Pet LR, Hsieh WH, Pencina MJ, Ward S, Pollack MH, Fava M. Efficacy of dose increase among nonresponders to low-dose aripiprazole augmentation in patients with inadequate response to antidepressant treatment: a randomized, double-blind, placebo-controlled, efficacy trial. J Clin Psychiatry. 2012 Mar;73(3):353-7. doi: 10.4088/JCP.10m06541. Epub 2011 Sep 20. PMID 21939613
- See also: A double-blind, placebo-controlled study of aripiprazole adjunctive to antidepressant therapy among depressed outpatients with inadequate response to prior antidepressant therapy (ADAPT-A Study) — https://www.ncbi.nlm.nih.gov/pubmed/22286203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 U.S. sites enrolled 225 patients over 10 months. 221 patients are included in the analysis. Enrollment began in September, 2008 and completed in July, 2009.
Pre-assignment Details: Patients completed a SAFER interview before randomization. No other significant events occurred prior to randomization.
Groups:
- ADAPT Drug/Drug Group: Patients randomly assigned to the drug/drug sequence: the dose of aripiprazole will be 2 mg/day during the first phase of the study, and 5 mg/day in the second phase.
- ADAPT Placebo/Placebo Group: Patients randomly assigned to the placebo/placebo sequence: the patients will receive a placebo treatment during the first phase of the study, and a placebo treatment in the second phase.
- ADAPT Placebo/Drug Group: Patients will be randomly assigned to placebo during the first phase of the study. In the second phase of the study, they will receive the aripiprazole drug at a dose of 2 mg/day.
Period: 30-Day Phase 1 Period
Arm/Group | ADAPT Drug/Drug Group | ADAPT Placebo/Placebo Group | ADAPT Placebo/Drug Group
Started | 56 | 84 | 85
Completed | 54 | 83 | 84
Not Completed | 2 | 1 | 1
Period: 30-Day Phase 2 Period
Arm/Group | ADAPT Drug/Drug Group | ADAPT Placebo/Placebo Group | ADAPT Placebo/Drug Group
Started | 54 | 83 | 84
Completed | 48 | 78 | 75
Not Completed | 6 | 5 | 9

BASELINE CHARACTERISTICS:
Population: This data was analyzed for the study by comparing placebo vs. drug. Therefore the two groups (placebo/placebo and placebo/drug) that started with placebo during the first phase of the study are combined as one group called Placebo. The patients who were took the study drug in both phases are in the Drug/Drug group.
Groups:
- ADAPT Drug/Drug Group: patients randomly assigned to the drug/drug sequence, the dose of aripiprazole will be 2 mg/day during the first phase of the study, and 5 mg/day in the second phase.
- ADAPT Placebo Group (Placebo/Placebo & Placebo/Drug Groups): This data was analyzed for the study by comparing placebo vs. drug. Therefore the two groups (placebo/placebo and placebo/drug) that started with placebo during the first phase of the study are combined as one group. Patients in the placebo/placebo sequence received a placebo treatment during the first phase of the study, and a placebo treatment in the second phase. Patients in the placebo/drug sequence received a placebo treatment during the first phase of the study and they received the aripiprazole drug at a dose of 2 mg/day in the second phase of the study.
- Total: Total of all reporting groups
Arm/Group | ADAPT Drug/Drug Group | ADAPT Placebo Group (Placebo/Placebo & Placebo/Drug Groups) | Total
Number analyzed (Participants) | 56 | 169 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 169 | 225
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.36 (10.35) | 45.06 (11.34) | 45.16 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 108 | 145
  Male | 19 | 61 | 80
Region of Enrollment [Number; unit: participants]
  United States | 56 | 169 | 225

OUTCOME MEASURES:

1. Primary Outcome: MADRS (Montgomery-Asberg Depression Rating Scale) Response Rate
Description: The primary outcome was the difference in response rate (decrease in MADRS total score of at least 50%) using the SPCD (sequential parallel comparison design). The 10-item Montgomery-Asberg Depression Rating Scale (MADRS), which measures depression severity over the past week, was completed by clinicians using an MGH structured interview. Each item is measured on a scale from 0 to 6, and the items are summed to find the total score. The total minimum score is 0 units on a scale and the total maximum score is 60 units on a scale, where higher scores indicate more severe depression.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Drug: Patients who received drug in phase 1 (aripiprazole 2 mg/day)
- Phase 1 Placebo Non-Responders on Drug in Phase 2: Patients who received (and had no response) to a Placebo in Phase 1 and then received drug (aripiprazole 2mg/day) in Phase 2
- Phase I Placebo: Patients who received Placebo in Phase 1
- Phase 1 Placebo Non-Responders on Placebo in Phase 2: Patients who received (and had no response) to a Placebo in Phase 1 and then received a placebo treatment in Phase 2
Arm/Group | Phase 1 Drug | Phase 1 Placebo Non-Responders on Drug in Phase 2 | Phase I Placebo | Phase 1 Placebo Non-Responders on Placebo in Phase 2
Number analyzed (Participants) | 54 | 61 | 167 | 63
Participants | 10 | 11 | 29 | 5

2. Secondary Outcome: MADRS (Montgomery-Asberg Depression Rating Scale) Readmission Rate
Description: MADRS readmission rate is defined as MADRS score<11. The 10-item Montgomery-Asberg Depression Rating Scale (MADRS), which measures depression severity over the past week, was completed by clinicians using an MGH structured interview. Each item is measured on a scale from 0 to 6, and the items are summed to find the total score. The total minimum score is 0 units on a scale and the total maximum score is 60 units on a scale, where higher scores indicate more severe depression.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Drug | Phase 1 Placebo Non-Responders on Drug in Phase 2 | Phase I Placebo | Phase 1 Placebo Non-Responders on Placebo in Phase 2
Number analyzed (Participants) | 54 | 61 | 167 | 63
Participants | 4 | 8 | 16 | 4

3. Secondary Outcome: Mean Change in MADRS (Montgomery-Asberg Depression Rating Scale) Score From Baseline to the End of Follow-up
Description: The 10-item Montgomery-Asberg Depression Rating Scale (MADRS), which measures depression severity over the past week, was completed by clinicians using an MGH structured interview. Each item is measured on a scale from 0 to 6, and the items are summed to find the total score. The total minimum score is 0 units on a scale and the total maximum score is 60 units on a scale, where higher scores indicate more severe depression.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 1 Drug | Phase 1 Placebo Non-Responders on Drug in Phase 2 | Phase I Placebo | Phase 1 Placebo Non-Responders on Placebo in Phase 2
Number analyzed (Participants) | 54 | 61 | 167 | 63
units on a scale | -8.54 (7.21) | -5.80 (7.08) | -8.09 (8.13) | -3.32 (5.97)

4. Secondary Outcome: Mean Change in Clinical Global Impression of Severity (CGI-S)
Description: The CGI-S scale was administered by clinicians based on assessment of the patient's clinical status. They measured, based on history and scores on other instruments, depressive severity. It consists of one question scored on a seven-point scale (1 = normal to 7 = among the most severe), so a higher total score indicates greater depressive severity. The minimum score is 1, and the maximum score is 7.
Time Frame: Baseline and 12 weeks
Population: This analysis used observed cases rather than LOCF (last observation carried forward), so some participants were missing follow-up data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 1 Drug | Phase 1 Placebo Non-Responders on Drug in Phase 2 | Phase I Placebo | Phase 1 Placebo Non-Responders on Placebo in Phase 2
Number analyzed (Participants) | 52 | 58 | 162 | 61
units on a scale | -0.81 (1.03) | -0.64 (0.95) | -0.84 (1.15) | -0.43 (0.78)

5. Secondary Outcome: Mean Change in Symptom Questionnaire (SQ)
Description: The SQ, a 92-item (yes/no) self-rating questionnaire, includes 4 distress and 4 well-being subscales. There are 68 items for the distress subscales and 24 items for the well-being subscales. Each item has either a Yes/No or True/False answer. For the distress symptom score, add together the following items and score 1 when the answer is Yes/True: 1, 2, 3, 5, 6, 8, 11, 12, 15, 18, 20, 22, 24, 25, 26, 27, 28, 29, 30, 32, 33, 34, 36, 37, 39, 41, 42, 44, 45, 47, 48, 49, 52, 53, 54, 55, 56, 57, 58, 59, 60, 61, 62, 63, 64, 65, 66, 67, 68, 69, 72, 73, 74, 75, 76, 77, 79, 80, 81, 82, 84, 85, 86, 87, 88, 90, 91, 92. Minimum score is 0 and maximum score is 68. A higher score indicates more distress symptoms. For the well-being subscale score, add together the following items and score 1 when the answer is No/False: 4, 7, 9, 10, 13, 14, 16, 17, 19, 21, 23, 29, 31, 35, 38, 40, 43, 46, 50, 51, 71, 78, 83, 89. Minimum score is 0 and maximum score is 24. A higher score indicates more well-being.
Time Frame: Baseline and 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 1 Drug | Phase 1 Placebo Non-Responders on Drug in Phase 2 | Phase I Placebo | Phase 1 Placebo Non-Responders on Placebo in Phase 2
Number analyzed (Participants) | 52 | 59 | 162 | 61
units on a scale
  Sum of 4 subscaled distress scores | -9.44 (11.19) | -6.78 (13.78) | -9.70 (12.51) | -4.52 (9.52)
  Sum of 4 subscaled well-being scores | 3.71 (5.12) | 3.34 (5.79) | 2.75 (5.88) | 1.98 (4.97)

6. Other Pre Specified Outcome: Treatment Emergent AEs in Two Treatment Groups - Safety Sample
Description: Differences in the incidence of treatment emergent AEs between the treatment groups were examined and evaluated using descriptive statistics. In this analysis, AEs were summarized according to person-phase of occurrence. Each AE was attributed to the person and then to phase 1 or phase 2, depending on the initial date of onset.
Time Frame: 12 Weeks
Population: AEs were summarized according to person-phase of occurrence. Each AE will be attributed to the person and then to phase 1 or phase 2, depending on the initial date of onset. If the severity or other characteristic of the AE changes between phases, it can be counted in both phases. Also see Table 5 in Reference.
Measure: Number; unit: adverse events
Units Other Than Participants: participant-phases
Groups:
- ADAPT Drug Group: Aripiprazole patient-phases from the Drug/Drug and Placebo/Drug Groups
- ADAPT Placebo Group: Placebo patient-phases from Placebo/Placebo and Placebo/Drug groups.
Arm/Group | ADAPT Drug Group | ADAPT Placebo Group
Number analyzed (Participants) | 115 | 167
Number analyzed (participant-phases) | 115 | 231
adverse events | 58 | 110

7. Other Pre Specified Outcome: Number of Patients With Treatment Emergent AEs in Two Treatment Groups - Placebo Non-Responders
Description: Differences in the incidence of treatment emergent AEs between the treatment groups were examined and evaluated using descriptive statistics. This analysis focused on placebo non-responders in phase 1 and presented them by their treatment assignment in phase 2.
Time Frame: 12 Weeks
Population: Of the 138 phase 1 placebo non-responders, 14 dropped out in phase 2: 9 in the drug arm and 5 in the placebo arm. Therefore, 124 total placebo non-responders from phase 1 were included in the analysis.
Measure: Number; unit: Patients
Arm/Group | Phase 1 Placebo Non-Responders on Drug in Phase 2 | Phase 1 Placebo Non-Responders on Placebo in Phase 2
Number analyzed (Participants) | 61 | 63
Patients | 40 | 44

8. Other Pre Specified Outcome: Number of Patients With Treatment Emergent AEs in Two Treatment Groups - People Exclusively on Drug or Placebo Throughout the Study
Description: Differences in the incidence of treatment emergent AEs between the treatment groups were examined and evaluated using descriptive statistics. This analysis compared AEs between the arms that received exclusively drug throughout the study or placebo throughout the study.
Time Frame: 12 Weeks
Measure: Number; unit: Patients
Groups:
- ADAPT Placebo/Placebo Group: Patients in the placebo/placebo sequence received a placebo treatment during the first phase of the study, and a placebo treatment in the second phase.
Arm/Group | ADAPT Drug/Drug Group | ADAPT Placebo/Placebo Group
Number analyzed (Participants) | 54 | 83
Patients | 39 | 60

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the 12 week study period.
Groups:
- Drug/Drug Group: Aripiprazole will be 2 mg/day during the first phase of the study, and 5 mg/day in the second phase for drug/drug group.
- Placebo/Placebo Group: Patients on placebo in phases 1 and 2
- Placebo/Drug Group: Patients on placebo in Phase 1 who are on drug in phase 2 (Aripiprazole 2 mg/day)
Arm/Group | Drug/Drug Group | Placebo/Placebo Group | Placebo/Drug Group
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/83 | 0/85
Other Adverse Events (participants affected / at risk) | 39/54 | 60/83 | 58/85
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Drug/Drug Group (N=54) | Placebo/Placebo Group (N=83) | Placebo/Drug Group (N=85)
Constipation (Gastrointestinal disorders) | 6 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 7 | 9
Nausea (Gastrointestinal disorders) | 5 | 9 | 4
Insomnia (Psychiatric disorders) | 5 | 7 | 7
Somnolence (Nervous system disorders) | 4 | 3 | 1
Fatigue (General disorders) | 3 | 1 | 5
Weight increased (Investigations) | 13 | 23 | 6
Headache (Nervous system disorders) | 4 | 9 | 13
Dry mouth (Gastrointestinal disorders) | 4 | 3 | 2
Oedema peripheral (General disorders) | 14 | 11 | 1
Nasopharyngitis (Infections and infestations) | 7 | 1 | 4
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less